CLINICAL TRIAL: NCT06915909
Title: Robotic Prostatectomy Artificial Intelligence Low Pressure Pain Study Trial - "The Monitoring of Patients Outcomes Intraoperatively and Perioperatively Using the Airseal and Stryker Insufflator Undergoing Robotic Assisted Laparoscopic Prostatectomy at a Pressure and Stability of Pneumoperitoneum of 8 mmHg"
Brief Title: Robotic Prostatectomy Artificial Intelligence Low Pressure Pain (RALP) Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD2024-75; 346481 (Other: IRAS (Integrated Research Application System) Project ID)
Record Dates: First submitted 2025-02-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Cancer (Post Prostatectomy); Prostate Cancer Surgery; Prostate Cancers; Prostate Neoplasm; Prostatectomy
Keywords: prostate cancer; prostatectomy; robotic prostatectomy; post-operative pain; pain; Stryker PneumoClear insufflator; AirSeal Insufflation System; intra-operative pain; Medasense
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Pain, Postoperative; Pain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, open label, human clinical study designed to evaluate pain related to the use of the AirSeal® Insufflation System (AIS) vs a Stryker PneumoClear Insufflator for the management of pneumoperitoneum.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stryker PneumoClear insufflator (Active Comparator): Measuring patient's pain during and after a robotic prostatectomy using the Stryker PneumoClear insufflator. 20 patients will be randomised and assigned to this arm of the trial. Post-op pain outcomes will be compared to the control arm (standard of care), the AirSeal Insufflation System.
  Interventions: Device: surgery
- AirSeal® Insufflation System (No Intervention): Measuring patient's pain during and after a robotic prostatectomy using the AirSeal® Insufflation System. 20 patients will be randomised and assigned to this arm of the trial. This device is the standard of care at the Lister hospital, Stevenage, UK.

INTERVENTIONS:
Device: surgery — 40 patients randomised to two arms will undergo robotic prostatectomies using either the control AirSeal® Insufflation System (AIS) or the intervention Stryker PneumoClear Insufflator. Intra-operative and post-operative pain will be compared between the two arms of the trial.
  Other Names: Robotic assisted laparoscopic prostatectomy
  Arms: Stryker PneumoClear insufflator

SUMMARY:
The 'Robotic Prostatectomy Artificial Intelligence Low Pressure Pain Study Trial' aims to assess the feasibility of being able to review operative outcomes such as pain when comparing two commonly used surgical devices for the removal of prostate cancers. The data collected will inform methodologies for future, larger, multi-center trials investigating pain in patients undergoing prostate cancer surgery.

A robotic prostatectomy is a commonly performed surgery used to treat prostate cancer by removing the prostate gland. In order to perform the procedure, the surgeon must 'inflate' (technical term pneumoperitoneum) the patients abdomen with carbon dioxide gas using a device called an insufflator. Adequate 'inflation' of the abdomen ensures the surgeon can clearly visualise the prostate. Unfortunately, higher pressures of abdominal 'inflation' are a large contributor to intra and post-operative pain in patients having prostatectomies. The type of insufflator device used to maintain inflation pressures in the abdomen are thought to be a variable contributing to differing levels of intra and post-operative pain. Therefore, the purpose of this trial is to compare intra and post-operative pain when using two different insufflator devices when performing robotic prostatectomies. Both insufflators are already commonly used across multiple NHS Trusts.

40 patients awaiting a robotic prostatectomy at the urology department at the Lister hospital, Stevenage, will be randomised to use either the Conventional Insufflator System (CIS) {Stryker PneumoClear Insufflator} or the AIRSEAL® Insufflation System (AIS) to 'inflate' their abdomens during their prostatectomies. Data relating to various intra and post-operative outcomes will be collected in the 30 days following the patient's operation. Outcomes include levels of intra and post-operative pain, medication use, procedure time, recovery room time, length of hospital stay, post operative nausea and vomiting and adverse events. This data can be analysed to identify trends in differences in outcomes between the AIS and CIS insufflators.

DETAILED DESCRIPTION:
In this trial, 40 patients undergoing robotic prostatectomies will be randomised to have either the AIRSEAL® Insufflation System (AIS) or the Stryker PneumoClear Insufflator devices used to maintain pneumoperitoneum during surgery. Data relating to intra-operative and post-operative pain will be collected. This data will be used to identify any differences in outcomes between the two arms of the trial.

The main aim of this feasibility study will be to inform the feasibility and design of a subsequent definitive full-scale trial. The feasibility trial will collect data about recruitment, study conduct, and assessment methods. The objectives of the feasibility are to

* Assess recruitment rates
* Evaluate whether the study can run in line with the study protocol
* Identify the feasibility of collecting clinical data
* Evaluate treatment-based adverse events, serious adverse events, anticipated adverse device effects, unanticipated adverse device effects and all device deficiencies and use errors, regardless of relationship to an adverse event
* Estimate the likely magnitude of the effect of the intervention. To allow for estimation of the sample size for the full trial

The subsequent large scale, multi-center trial following this feasibility trial will focus on severity of pain during and immediately after surgery in the recovery room and then by 6-hour increments, measured by a 0 - 10 Numeric Rating Scale (NRS) and a PMD-200 nociception non-invasive monitor as the primary outcome

Secondary outcomes include:

Pre-Operative

1. Pre-op vitals including height and weight
2. Pre-op labs

Intra-operative

1. Insufflation Pressure
2. Estimated blood loss
3. Blood transfusion (intra-operative)
4. Procedure time (initial incision to closure)
5. Surgeon-determined need to increase IAP beyond "study pressure"
6. Administration of transversus abdominis plane block
7. Urine output
8. Anesthetic/pain medication administration
9. MedaSense PMD-200 monitor for pain documentation
10. Intraoperative Peak Airway Pressure every 15 minutes
11. Intraoperative End Tidal Carbon Dioxide (ETCO2) every 15 minutes

Post-Operative During hospital discharge, all subjects will be evaluated for incidence and severity of pain using a 0-10 numeric rating scale (NRS) and records of medication use and a PMD-200 monitor. These data will be captured in the Case Report Forms.

Recovery room:

1. Time in recovery room
2. Post-op pain incidence and severity (abdominal) NRS
3. Pain medications
4. Post- op labs (CBC, Chem-7) per standard of care
5. Vital signs 24 hr

Discharge:

1. Post-op pain incidence and severity (abdominal) NRS
2. Presence or absence of postoperative nausea or vomiting
3. Pain medications
4. Length of hospital stay
5. Pain Interference and Pain Intensity short form surveys
6. Any complications that were observed. Post-operative complications through 30 days, reported using Clavien-Dindo Classification, including 30-day mortality
7. Return to operating room within 24 hour
8. Readmission to hospital within 30 days

Classification, including 30-day mortality

All Adverse Events (intra-operative and post-operative through 30 days):

1. Adverse Events
2. Serious Adverse Events
3. Anticipated Adverse Device Effects
4. Unanticipated Adverse Device Effects 5 All device deficiencies and use errors, regardless of relationship to an adverse event

Patients under the care of the urology department at the Lister Hospital, Stevenage will be listed in clinic for a robotic prostatectomy. If patients meet the eligibility criteria for the trial, they will be approached and informed of the RALP clinical trial during their clinic consultation, by a member of the clinical team (likely a urological consultant).

Patients will be provided with a patient information sheet informing them of the aims and methodology of the trial. Members of the research department will be able to answer any outstanding questions patients might have.

Written informed consent will be obtained from eligible patients (n=40) willing to participate in the trial. If patients consent, their GP will subsequently be written to and informed of their involvement in the trial.

Pre-Operative data collection:

Within 30 days of a subject's scheduled procedure, members of the research department at Lister hospital will obtain a medical history and record the subject's demographic (age, race, sex and date of birth) and baseline information (height, weight, and systolic/diastolic blood pressure). Within 30 days prior to the planned procedure date, obtain serum blood tests per standard of care. These will typically include:

• FBC • Renal function test • CRP This data, along with all subsequent trial related data will be anonymised and subsequently inputted into a database created by the Centre for Health Services and Clinical Research at the University of Hertfordshire.

Preoperative Randomization:

Randomization will be done electronically via a database which is facilitated by the University of Hertfordshire. Patients will be randomized 1:1 to either AIS (at 8 mmHg) or Stryker PneumoClear Insufflator Arm 1: AIRSEAL® Insufflation System (AIS) - 8 mmHg Arm 2: Stryker PneumoClear Insufflator - 8 mmHg.

Methods and Procedure:

Patients will undergo their robotic assisted prostatectomy with the use of either the AIRSEAL® Insufflation System (AIS) or Stryker PneumoClear Insufflator depending on which arm of the trial they have been randomized to. Patients will be blinded to the intervention (AIRSEAL® Insufflation System (AIS) or Stryker PneumoClear Insufflator). Both systems are commonly used devices across many NHS trusts and there is currently no evidence comparing patient outcomes between use of the two devices.

This study will be conducted at one site by one surgeon performing 40 total procedures. Study subjects will be prepared for surgery per standard institutional policy and practice. Standard operative procedures will be followed.

Case Report Forms will be also be used to collect data relating to pre-operative, intra-operative and post-operative outcomes. This data will relate to outcomes such as intra-operative pain, post operative pain scores, medication use, duration of hospital stay, presence of nausea or vomiting etc...

The final patient follow up will be in a clinic appointment 30 days following their operation. Ongoing post-operative outcomes will be assessed (pain scores, medication use, adverse events etc...).

Data will be inputted on the database which is subsequently processed and statistically analysed and reviewed. Differences in outcomes between the two arms of the trial may be identified.

Once the aforementioned data has been processed and reviewed, results may be published and also distributed to those trial participants who wished to receive ongoing information and results from the trial.

The outcomes of this research will be used to inform future research such as a full scale trial with a larger number of patients and larger volume of data

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for non-emergent robotic Prostatectomy surgery
* Patients (or appropriate legal representatives) able to provide written informed consent to participate in the study
* Males, aged 18 to 75 years
* Have no significant psychopathology that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioural recommendations and office visits
* Are American Society of Anaesthesiologists (ASA) Class I, II, or III);

Exclusion Criteria:

* Patient participation in a different investigational clinical study within 90 days before screening and for the duration of this trial (unless previously approved by the investigator and Sponsor);
* Patients requiring any surgical procedure in addition to Prostatectomy and or / Pelvic Lymph node dissection
* Previous pelvic surgery or previous malabsobtion or restrictive procedures performed for the treatment of obesity
* Inability to provide informed consent
* Unable or unwilling to attend follow-up visits and examinations
* Uncontrolled hypertension (=/>Systolic: 180 mmHg/Diastolic: 120 mmHg) and/or diabetes mellitus (Blood sugar level: >200 mg/dL)
* Patients who fall into American Society of Anesthesiologists (ASA) Class ≥ IV
* History of chronic alcohol or drug abuse within 2 years of the screening visit
* Chronic renal failure or on dialysis
* Significant complicating medical history or immunocompromised
* History or presence of pre-existing autoimmune connective tissue disease, e.g., systemic lupus erythematosus or scleroderma
* Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
* Any medical condition which precludes compliance with the study
* Subjects with any other clinically significant unstable medical disorder, life threatening disease, or conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study or which would contra-indicate a surgical procedure.
* Previous or current history of being on regular analgesia / pain killers

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | Through study completion estimated to be 6-12 months
Evaluate treatment-based adverse events, serious adverse events, anticipated adverse device effects, unanticipated adverse device effects and all device deficiencies and use errors, regardless of relationship to an adverse event. | Through study completion estimated to be 6-12 months
Pre-op vitals | Baseline/day 1
  Bloods pressure, heart rate, oxygen saturations, respiration rate, temperature
Pre-op BMI (height and weight) | Baseline/day 1
  kg/m^2
Pre-op labs | Baseline/day 1
  Pre-op FBC, U&E, CRP and PSA bloods
Insufflation Pressure | Perioperative
  Intraoperative insufflation pressure (mmHg)
Estimated blood loss | Perioperative
  Estimated intra-operative blood loss (ml)
Blood transfusion | Perioperative
  Intra-operative blood transfusions (number of units of blood e.g 0, 1, 2, 3 etc...)
Procedure time (initial incision to closure) | Perioperative
  Number of minutes from incision to closure
Surgeon-determined need to increase IAP beyond "study pressure" | Perioperative
  Need to increase insufflation pressure intra-operatively (mmHg)
Administration of transversus abdominis plane block | Perioperative
  Was a transversus abdominis plane block administered (yes or no)
Anesthetic/pain medication administration | Perioperative
  Intra-operative administration of analgesia (morphine milligram equivalent units)
MedaSense PMD-200 monitor for pain documentation | Perioperative
  Intra-operative pain score (NOL score 0-100)
Intraoperative Peak Airway Pressure every 15 minutes | Perioperative
  Intra-operative PAP (cmH2O)
Intraoperative End Tidal Carbon Dioxide (ETCO2) every 15 minutes | Perioperative
  Intra-operative ETCO2 (mmHg)
Time in recovery room | Perioperative
  Number of minutes spent in post-op recovery
Post-op pain incidence and severity | Day 1-30 post-op/post-intervention
  Pain measured using visual analogue scale, numerical rating scale and pain incidence and interference surveys. Pain surveys done at 1, 3, 6, 12, 18, 24 hours and day 7 and day 30 post-operation.
Post-op analgesia usage | Day 1-30 post-op/post-intervention
  Post-op analgesia usage on discharge (morphine milligram equivalent units)
Post- op labs as per standard of care | Day 1-30 post-op/post-intervention
  FBC, U&E, CRP
Vital signs 24 hr | Day 1 post-op/post-intervention
  Blood pressure, heart rate, respiration rate, oxygen saturations, temperature
Presence or absence of postoperative nausea or vomiting | Day 1 post-op/post-intervention
  Presence of nausea/vomiting in the post-op period
Length of hospital stay | Day 1-30 post-op/post-intervention
  Duration of hospital admission (hours)
Any complications that were observed. Post-operative complications through 30 days, reported using Clavien-Dindo Classification, including 30-day mortality | Day 1-30 post-op/post-intervention
  Reporting of post-operative complications
Return to operating room within 24 hour | Day 1-30 post-op/post-intervention
  Reason for return to the operating room and number of returns to operating room
Readmission to hospital within 30 days | Day 1-30 post-op/post-intervention
  Reason and number of readmissions to hospital
All Adverse Events (intra-operative and post-operative through 30 days) | Day 1-30 post-op/post-intervention
  Documented using the "Common Terminology Criteria for Adverse Events" (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Lister hospital, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT06915909/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT06915909/SAP_001.pdf
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT06915909/ICF_002.pdf